CLINICAL TRIAL: NCT00836238
Title: A Cross-Sectional Study of the Predictability of a Questionnaire About Difficulty in Climbing Up or Down Stairs in Objective Measures of Functional Status in Elderly Patients With Prostate Cancer
Brief Title: Questionnaire and Fall Risk Assessment
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2008-0779
Record Dates: First submitted 2009-01-26; First posted 2009-02-04 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Neural Functioning Assessment; Physical Assessment; Questionnaire; Objective Measures of Functional Status; Physical Function; Symptom Assessment Interview; Elderly
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Interviews as Topic; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Questionnaire + Fall Risk Assessment: Physical Function Interview + Physical Function Tests + Symptom Assessment Interview
  Interventions: Behavioral: Interview; Other: Physical Function Tests

INTERVENTIONS:
Behavioral: Interview — Physical Function and Symptom Assessment Interviews
  Other Names: survey
Other: Physical Function Tests — 3 physical function tests.

SUMMARY:
The goal of this research study is to learn if your answers to questions during an interview can help researchers predict how well you function physically and if you are at a high risk for falls.

Primary Objectives:

-To determine how accurately a simple questionnaire can predict three objective measures of function in elderly patients with prostate cancer.

Secondary Objectives:

* To assess the correlations between three functional tests and the number of self-reported falls in elderly patients with prostate cancer.
* To determine risk factors related to number of falls in elderly prostate cancer patients.

DETAILED DESCRIPTION:
Physical Function Interview:

If you agree to take part in this study, you will be asked 6 questions. The first 2 questions ask about your physical ability to walk up and down stairs. The next 4 questions ask about your history of falling down in the last year, symptoms of depression, loss of urinary control, vision problems, and your ability to function physically. If you report that you have fallen down more than 3 times in the last year, you will automatically be referred for a physical therapy evaluation at M. D. Anderson.

Physical Function Tests:

After you have completed the questionnaires, you will perform 3 physical function tests:

* For the first test, you will sit in a chair, stand up, walk 10 feet as quickly and safely as possible, turn around, return to the chair and sit again. This test will be timed. You will perform this test 3 times, the average of the times will be recorded. There will be no rest break between each test.
* For the next test, you will stand only on 1 leg as long as possible, and this time will be recorded.
* You will complete a grip strength test. You will grip a small device in 1 hand and squeeze as hard as you can while you are in a seated position. You will perform this test 3 times and your best measurement will be recorded. There will be no rest period between the 3 tests.

Symptom Assessment Interview:

After you complete the physical function tests, you will be asked to rate any symptoms you experience on a scale from 0-10 (with 0 being the best and 10 being worst). You will be asked to rate symptoms of things such as pain, fatigue, nausea, depression, anxiety, drowsiness, and shortness of breath.

Medical Record Information:

Information will be collected from your medical record. This information will include your age, race, gender, weight, height, body mass index, disease diagnosis, history of chemotherapy and medications, and medical history.

Additional Information:

The physical function interview, tests of physical function, and symptom assessment interview will take about 45 minutes total to complete during an already-scheduled visit to the clinic.

Length of Study:

Your participation on this study will be over after you have completed the questionnaires, physical function tests, and the symptom assessment.

This is an investigational study. Up to 60 people will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have the ability to understand and willingness to sign a written informed consent document.
2. Patients must be able to ambulate with or without an assistive device, without assistance from a person.
3. Patients must be 65 years old or older.
4. Patients must have a diagnosis of prostate cancer
5. Patients must have received androgen deprivation therapy (ADT) for their prostate cancer for at least 3 months and were responding to treatment as determined by prostate-specific antigen criteria.
6. Patients have received chemotherapy within last month.
7. Patients must speak English.

Exclusion Criteria:

1. Patients who decline to participate or who are determined incapable of completing the study.
2. Active Central Nervous System (CNS) disease such as clinically-evident CNS metastases or leptomeningeal disease, dementia, or encephalopathy (per treating physician's assessment).

Min Age: 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Males with prostate cancer, 65 years of age or older, who able to ambulate with or without an assistive device, without assistance from a person.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2009-02; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Number Patient Falls + Activity Limitations Using Functional Tests | 45 minutes total to complete during already-scheduled clinic visit

CONTACTS AND LOCATIONS:
Overall Officials: Ying Guo, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org